CLINICAL TRIAL: NCT00941265
Title: Effect of Dopaminergic Medication on Recovery of Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Leemann Beatrice, Dr., University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 05-159 (NAC 05.051)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Aphasia
Keywords: treatment of anomia; levodopa; patient with aphasia hospitalised at the "Service de neurorehabilitation" with presence of anomia
MeSH Terms: conditions — Aphasia | interventions — benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levodopa 100 mg and benserazide 25 mg (Other): 2 weeks with Daily CAT on list A+ levodopa and benserazide
  Interventions: Drug: levodopa and benserazide
- placebo (Other): 2 weeks with Daily CAT on list B + placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levodopa and benserazide — Daily Monday to Friday CAT with Daily Monday to Friday levodopa 100 mg with benserazide 25 mg , in the morning 1 h after breakfast, during 2 weeks .
  Arms: levodopa 100 mg and benserazide 25 mg
Drug: placebo — Daily CAT Monday to Friday with daily placebo Monday to Friday , in the morning 1 h after breakfast, taken 5 out of 7 days during the 2 weeks of one of the two treatment periods.
  Arms: placebo

SUMMARY:
The investigators have been offering computer assisted therapy of aphasia (CAT) as a complement to traditional treatments to aphasia patients of the "Service of Neurorehabilitation" for some years. The investigators have shown its efficacy in hospitalised patients with recently acquired aphasia.

In addition to studies stressing the importance of treatment intensity, several studies suggest that pharmacological treatment can also improve recovery after a cerebral lesion. The underlying idea is that the administration of medication influencing the system of neurotransmitters can play a role in functional recovery. Studies have assessed mainly substances acting on the dopaminergic (amphetamine and bromocriptine) and GABAergic system (piracetam).

The main objective of the present study concerns the evaluation of the effects of levodopa on recovery of anomia in patients with aphasia. In particular, the investigators use CAT to control intensity and quality of therapy and they will assess whether the administration of levodopa promotes recovery.

In each patient, two periods of anomia therapy with CAT, each performed with a different word list, will be compared. In addition to speech therapy, each period will be associated with the administration of either levodopa and benserazide (Madopar ®), or placebo. Evaluations at baseline and after each treatment period will be performed with the material and denomination battery

ELIGIBILITY:
Inclusion Criteria:

* Patient with aphasia hospitalised at the "Service of neurorehabilitation" with presence of anomia absence of comprehension deficits, absence of executive or apraxic dysfunctions that might impede the handling of keyboard or mouse, absence of stereotypies or perseverations dominating the aphasic symptoms.

Exclusion Criteria:

* Patients who do not have their ability to judge or who suffer from Parkinson's syndrome requiring dopaminergic treatment will be excluded. Moreover, absolute medical contraindications for the medication will be respected: known hypersensitivity to one of the components, patients taking MAO inhibitors or sympathomimetics, severe hormonal, renal, hepatic, or cardiac affections, pregnancy or breastfeeding, women at reproductive age without reliable contraception, angle closure glaucoma, psychosis or severe neurosis, age < 25 years, malign melanoma, or planned anesthesia during the study period + 48 hours.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
performance in denomination in the two word list will be compared | at the begining , at two weeks and at 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Armin Schniider, Prof, Study Director — University Hospital, Geneva
Locations (1):
- Neurorééducation, University Hospital, Geneva, Switzerland